CLINICAL TRIAL: NCT03395860
Title: Low Dose Rabbit Antithymocyte Globulin Plus Low-dose Post-transplantation Cyclophosphamide as GVHD in Hapl-HSCT for Patients With Hematologic Malignancies: a Phase II Trial
Brief Title: Low Dose ATG Plus Low Dose PTCy as GVHD Prophylaxis in Haplo-HSCT
Acronym: ATG/PTCy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Head of Hematology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-ATG/PTCy; NSFC (Other Grant/Funding Number: 81370601)
Record Dates: First submitted 2017-12-30; First posted 2018-01-10 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2018-05

CONDITIONS: Graft-versus-host-disease; Prophylaxis
Keywords: GVHD; ATG; PTCy; halo-HSCT
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Intervention Model Description: drug: rATG drug: PTCy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): low dose antithymocyte globulin rATG(2.5mg/kg/d) used at d-3-d-2 low dose post-transplant cyclophosphamide PTCy (50mg/kg/d) use at d+3
  Interventions: Drug: ATG
- group B (Experimental): low dose antithymocyte globulin rATG(2.5mg/kg/d) used at d-2-d-1 low dose post-transplant cyclophosphamide PTCy (50mg/kg/d) use at d+3
  Interventions: Drug: ATG

INTERVENTIONS:
Drug: ATG — group A:low dose antithymocyte globulin rATG(2.5mg/kg/d) used at d-3-d-2 low dose post-transplant cyclophosphamide PTCy (50mg/kg/d) use at d+3 group B:low dose antithymocyte globulin rATG(2.5mg/kg/d) used at d-2-d-1 low dose post-transplant cyclophosphamide PTCy (50mg/kg/d) use at d+3
  Other Names: PTCY

SUMMARY:
Low dose Rabbit Antithymocyte Globulin plus Low-dose post-transplantation cyclophosphamide as graft-versus-host disease prophylaxis in haploidentical hematopoietic stem cell transplantation for patients with hematologic malignancies

DETAILED DESCRIPTION:
A novel regimen, which is composed of a low dose of ATG (5 mg/kg) and low-dose PTCy (one dose of PTCy, 50mg/kg) for GVHD prophylaxis in haplo-HSCT for patients with hematologic malignancies, is going to be evaluated in the prospective, randomized control, phase II clinical trial. It is theoretically feasible because the mechanisms of ATG and Cyclophosphamide on T lymphocyte are different. ATG plays the immunosuppressive activity on the depletion of peripheral T lymphocytes through complement dependent lysis or activation-associated apoptosis. ATG also modulates cell-surface expression of surface adhesion molecules or chemokine receptors. In addition, ATG can also affect or interfere with the function of different immune cells such as B lymphocytes, regulatory T lymphocytes (Treg), natural killer (NK)-T lymphocytes and dendritic cells (DC).Cyclophosphamide is nontoxic to hematopoietic stem cells and can selectively deplete the alloreactive T cells. Therefore, we hypothesis that ATG followed by PTCy have the synergistic effect on GVHD prophylaxis. (2) Luznik et al also showed that there was no difference in the incidence of severe acute GVHD between one or two doses of PTCy. Furthermore, there was a trend toward a lower incidence of extensive cGVHD among patients of two doses of PTCy compared with one dose PTCy. One dose of PTCy might preserve the GVL effect without influencing the incidence of the severe aGVHD. (3) Y Wang et al reported a randomized clinical trial comparing two different doses of ATG (6 and 10mg/kg) as GVHD prophylaxis for Haplo-HSCT. There was no difference in the median myeloid and platelet engraftment time and the rate of graft failure. The results showed that the incidence of grade III-IV acute GVHD was higher in the ATG-6 group than in the ATG-10 group. But the EBV reactivation occurred more frequently in the ATG-10 group than in the ATG-6 group. The higher rate of infection and NRM may influence the transplant outcomes in this GVHD prophylaxis strategy. We speculated that low dose of ATG (5 mg/kg) will ensure the engraftment and decrease infection frequency. But the optimal timing of ATG administration still needed to be considered. The immunosuppressive activity of ATG is not only dose-dependent but also rely on the timing of drug administration, especially when the lower dose of ATG was used as GVHD Prophylaxis. So we designed a randomized control phase II study to evaluate the efficacy and toxicity with low dose ATG followed by low dose PTCy as GVHD prophylaxis .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hematologic malignancies (AML, ALL, high-risk MDS, lymphoma, CML) were enrolled in this study. Diagnosis was according to the criteria of 2008 World Health Organization (WHO) classification of tumors of hematopoietic and lymphoid tissues.
* Family members selected as donors were typed at the HLA-A, -B, -DQB1, -C and -DRB1 locus at high-resolution level. Haplo was defined as recipient-donor number of HLA mismatches > 2.(20)
* 14 to 70 years old.
* Performance status scores no more than 3 (ECOG criteria).
* Adequate organ function as defined by the following criteria: alanine transaminase （ALT）, aspartate transaminase（AST） and total serum bilirubin <2×ULN (upper limit of normal). Serum creatinine and blood urea nitrogen (BUN) <1.25×ULN.
* Adequate cardiac function without acute myocardial infarction, arrhythmia or atrioventricular block, heart failure, active rheumatic heart disease and cardiac dilatation(the patients has been improved after treatment of the disease and are not expected to affect transplant can include in the study).
* Absence of any other contraindications of stem cell transplantation. Willingness and ability to perform HSCT.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Presence of any condition inappropriate for HSCT.
* Life expectancy < 3 months because of other severe diseases.
* Presence of any fatal disease, including respiratory failure, heart failure, liver or kidney function failure.
* Uncontrolled infection.
* Pregnancy or breastfeeding.
* Has enrolled in another clinical trials.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidences of acute GVHD | 100 days after transplantation
  The cumulative incidences of aGvHD was defined as the number and the ratio of the participants with aGVHD

SECONDARY OUTCOMES:
Leukocyte engraftment | 1 MONTH
  Leukocyte engraftment:(was defined as the first of three consecutive days of peripheral white blood count >1000/ul.
Platelet engraftment | 1 MONTH
  Platelet engraftment:(was defined as the first of seven consecutive days of platelet counts of >50000/ul.
Donor chimerism | 2 YEARS
  Quantitative chimerism analyzes were performed using short-tandem-repeat-based polymerase chain reaction technique sat regular intervals for every 4 weeks after allografting in bone marrow.
Relapse incidence (RI) | 2 YEARS
  RI was defined as the number and ratio of the participants with relapse after transplantation
chronic GVHD | 2 year
  cGvHD was diagnosed and graded according to the 2014 National Institutes of Health (NIH) consensus criteria: mild, moderate or severe respectively.The number and ratio of participants with cGVHD after transplatation
infection | 6 month
  CMV and EB infections(The number and ration of participants with infection after transplantaton)

CONTACTS AND LOCATIONS:
Overall Officials: xinpeng wang, doctor, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai First People's HOSPITAL, Shanghai, Shanghai Municipality, China